CLINICAL TRIAL: NCT05924763
Title: The Clinical Outcome of the Biphasic Cartilage Repair Implant (BiCRI) in the Treatment of Chondral and Osteochondral Lesions of the Knee.
Brief Title: The Clinical Outcome of BiCRI in the Treatment of Chondral and Osteochondral Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioGend Therapeutics Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR18-001
Record Dates: First submitted 2023-05-25; First posted 2023-06-29 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2023-01

CONDITIONS: Articular Cartilage Disorder of Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BiCRI (Experimental): Biphasic Cartilage Repair Implant
  Interventions: Device: Biphasic Cartilage Repair Implant (BiCRI)

INTERVENTIONS:
Device: Biphasic Cartilage Repair Implant (BiCRI) — The Biphasic Cartilage Repair Implant (BiCRI) is a two-phase scaffold composed of poly(lactic-co-glycolic acid) (PLGA) and β-triCalcium phosphate (TCP).

SUMMARY:
Based on the previous successful experiences, the investigators like to extend our patient population. In this study, the investigators aim to determine the safety and effectiveness of the Biphasic Cartilage Repair Implant (BiCRI) in the treatment of chondral and osteochondral lesions of the knee, including but not limited to more than one (1) lesion and the lesion that had been treated with microfracture or mosaicplasty but failed.

DETAILED DESCRIPTION:
Patients who qualify for this trial and who are interested in participating will be consented using an Institutional Review Board (IRB) approved Informed Consent. Once a patient has signed the Informed Consent Form he/she is considered enrolled in the trial. If during surgery the size of lesion is found to meet exclusion criteria, the subject will be considered withdrawn (screen failure) from the trial.

Clinical trial eligibility should be determined by confirmation that the patient meets the criteria included in the Protocol. Standard arthroscopic technique should be used to fully assess the joint and determine if the chondral or osteochondral defect is appropriate for inclusion in the study. Through arthroscopic examination after initial debridement, the investigator should use his best judgment to estimate the size of the lesion, and the number of BiCRI to be applied.

Plain radiographs and MRI prior to 6-month (inclusive) visit will be performed according to routine clinical practice; however, 12-month and 24-monthpostoperative images should be done for study outcome evaluation

ELIGIBILITY:
Inclusion Criteria:

1. - Age between 16~65 (inclusive) years old presenting with either symptomatic chondral or osteochondral lesion of knee requiring primary surgical intervention. The lesions may include but not limited to following conditions:

   * multiple lesions
   * lesion that had been treated with microfracture or mosaicplasty but failed.
2. The index lesion is ICRS grade 3-4 lesion, Outerbridge grade 4, or OCD grades 3-4
3. Willing and able to consent in wiring to participate in the study

Exclusion Criteria:

* 1. Rheumatoid arthritis and other inflammatory arthritis 2. The index cartilage lesion requires more than 3 (exclusive) implants 3. Skeletally immature (epiphyses are not closed based on x-ray) 4. Concomitant comorbidities 5. Local or systemic infection, not including asymptomatic urinary tract infection if treated with antibiotics preoperatively 6. Pregnancy or breast feeding 7. Prisoner 8. Patient is actively participating in another medical device, drug, or biologic investigation (active defines as within the last 30 days prior to signing the consent form) 9. Any condition that is not suitable to participate in the study based on the physician's judgement

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-08-18 (Actual)

PRIMARY OUTCOMES:
International Knee Documentation Committee-2000 Subjective Knee Evaluation | 24 months after operation
  International Knee Documentation Committee-2000 Subjective Knee Evaluation compare to baseline
International Knee Documentation Committee-2000 Knee Examination Form | 24 months after operation
  International Knee Documentation CommitteeC-2000 Knee Examination Form compare to baseline
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 24 months after operation
  Knee Injury and Osteoarthritis Outcome Score (KOOS) compare to baseline
Pain (visual analogue scale;VAS) | 24 months after operation
  Pain (visual analogue scale;VAS) compare to baseline
Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) scale | 24 months after operation
  Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) scale

SECONDARY OUTCOMES:
International Knee Documentation Committee-2000 Subjective Knee Evaluation | 12 months after operation
  International Knee Documentation Committee-2000 Subjective Knee Evaluation compare to baseline
International Knee Documentation Committee-2000 Knee Examination Form | 12 months after operation
  International Knee Documentation CommitteeC-2000 Knee Examination Form compare to baseline
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 12 months after operation
  Knee Injury and Osteoarthritis Outcome Score (KOOS) compare to baseline
Pain (visual analogue scale;VAS) | 12 months after operation
  Pain (visual analogue scale;VAS) compare to baseline
Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) scale | 12 months after operation
  Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) scale

CONTACTS AND LOCATIONS:
Overall Officials: Gwen Chang, Study Director — BioGend Therapeutics Co.Ltd
Locations (2):
- Taiwan (2):
  - En Chu Kong Hospital, New Taipei City
  - Ministry of Health and Welfare Shuang-Ho Hospital, New Taipei City

IPD SHARING:
Plan to Share IPD: No